CLINICAL TRIAL: NCT07152392
Title: Evaluation of the Efficacy and Safety Observation of IBI311 Treatment in Patients With Inactive TAO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAP-3
Record Dates: First submitted 2025-06-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Associated Ophthalmopathies
Keywords: IGF-1R; TED; MR Imaging
MeSH Terms: conditions — Graves Ophthalmopathy; Insulin-Like Growth Factor I, Resistance To

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI311 (Active Comparator): Participants with inactive thyroid ophthalmopathy will 8 infusions of IBI1311 (10 mg/kg for the first infusion and 20 mg/kg for the remaining 7 infusions),The interval between each treatment is 3 weeks. After completing 4 treatments, observe for 3 months before entering the next stage of treatment。
  Interventions: Drug: IBI311
- Follow-up (Other): Participants with inactive thyroid ophthalmopathy will only receive follow-up every six months.
  Interventions: Other: Follew-up

INTERVENTIONS:
Drug: IBI311 — IBI311 is a fully human anti-IGF-1R mAb. IBI311 will be provided in single-dose 500-mg glass vials as a Injection solution containing.
  Arms: IBI311
Other: Follew-up — recived follow-up every six months
  Arms: Follow-up

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is an organ-specific autoimmune disease closely related to thyroid disease, which leads the incidence of orbital disease in adults and is the most common cause of diffuse toxic goiter (Graves disease, GD). The clinical manifestations of TAO are complex and varied. In severe cases, it may seriously impair visual function, affect daily life, and even cause corneal ulceration, perforation, and blindness. Therefore, a reasonable and effective treatment plan should be chosen according to the degree of TAO.

IBI311 is a fully human monoclonal insulin-like growth factor-1 receptor inhibitory antibody. It has binding activity against IGF-1R positive cells, can block the binding of IGF-1 and IGF-2 to IGF-1R, and has a dose-dependent effect. It can inhibit the proliferation of HT29 cells caused by the activation of the IGF-1R signaling pathway. Meanwhile, it can dose-dependently inhibit the proliferation of orbital fibroblasts and the secretion of hyaluronic acid (HA) in patients with TAO.

However, there are still significant gaps in the existing research evidence: There is a lack of reports on the efficacy and safety of IBI311 in inactive moderate to severe TAO patients.

The aim of this clinical study is to:

1. To evaluate the efficacy of IBI311 treatment in patients with inactive moderate to severe TAO.
2. To observe the safety of IBI311 treatment in patients with inactive moderate to severe TAO.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with TAO by Bartley criteria.
* Moderate to severe patients defined by EUGOGO.
* CAS <3 (on the 7-item scale) for the study eye.
* Participant with intractable diplopia, or incomplete closure of both eyes, or requiring further surgical intervention.
* Participant with a strong willingness for further intervention.

Exclusion Criteria:

* Anticipated need for intervention due to sight-threatening complications or other significant and acute deterioration in vision.
* Combined with other lesions in the orbit.
* Receive orbital radiotherapy or surgical treatment for TED, including orbital decompression, strabismus surgery and eyelid retraction correction.
* During the screening period, if either ear has a history of tinnitus or other hearing impairment; Or abnormal pure tone audiometry results (defined as an average bone conduction hearing threshold of ≥25 dB at 0.5, 1, 2, 4 kHz or a bone conduction hearing threshold of ≥40 dB at any frequency).
* At the time of screening, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times ULN, or accompanied by active hepatitis B (defined as HBsAg positive with HBV-DNA load greater than 1000 IU/ mL), or being receiving anti-hepatitis B virus treatment.
* During screening, the Glomerular Filtration Rate (GFR) was < 30 ml/ min/1.73m2 (using the MDRD formula: GFR =186× serum creatinine (mg/ dl) -1.154× (age) -0.203× (0.742 [if female]), unit conversion of serum creatinine: 1 μmol/L=0.0113 mg/dL); 10) At the time of screening, there was poorly controlled diabetes (defined as glycated hemoglobin ≥7.0% at the time of screening, or a new diabetes drug [oral or injection] or a dose change of the current prescribed diabetes drug > 10% within 60 days before screening).
* Screening for poorly controlled hypertension, with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; Or adjust the antihypertensive drug (dosage or type of drug) within 30 days before screening; Evidence of renal artery stenosis or unstable blood pressure (including orthostatic hypotension, etc.).
* At the time of screening, the 12-lead ECG showed a heart rate of < 50 beats/min or > 100 beats/min. The ECG indicated active heart disease, or the researchers believed that the abnormal ECG at the time of screening would interfere with the interpretation of the ECG results in the subsequent follow-up process. Especially, QTcF > 450 ms (for men) and QTcF > 470 ms (for women) should be excluded.
* HIV antibody or HCV antibody positive individuals or those with active syphilis (defined as those with positive non-specific syphilis antibodies or those who need anti-syphilis treatment after consultation by the infectious disease department).
* Any major illness/condition or evidence of an unstable clinical condition that, in the investigators judgment, will substantially increase the risk to the participant, or confound the interpretation of safety assessments, if they were to participate in the study.
* Any other condition that, in the opinion of the investigator, would impair the ability of the participant to comply with the study procedures or impair the ability to interpret data from the participants participation in the study.
* Pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2035-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were diplopia responders after 4 times and at the end of the treatment | up to 24 weeks
  Diplopia responders were defined as percentage of participants with ≥ 1 class improvement of eye motility from baseline assessed by Gorman score.
  Gorman score: 1 = no diplopia, 2 =intermittent diplopia, 3 = inconstant (gaze-evoked) diplopia, 4 = constant diplopia in primary or reading position.
Percentage of participants who were proptosis responders after 4 times and and the end of the treatment | up to 24 weeks
  Proptosis responders were defined as subjects whose exophthalmos in the study eye decreased by ≥2 mm compared to the baseline, and whose exophthalmos in the contralateral eye did not deteriorate (increase by ≥2 mm) at the end of the treatment.
Incidence and characterization of nonserious treatment emergent adverse events (TEAEs) during the treatment | throughout the study period

SECONDARY OUTCOMES:
Percentage of participants who were ATA categorical responders after 4 times and at the end of the treatment | up to 24 weeks
  Participants whose baseline ATA score of the study eye was >4, with a reduction of ≥1 grade in the ATA score, while there was no corresponding deterioration in the contralateral eye (≥1 grade deterioration).
  The denominator is the number of subjects with a baseline ATA score grade >4.
Change of GO-QoL from baseline after 4 times and at the end of the treatment | up to 24 weeks
Changes of the visual field in the dark areas from baseline after 4 times and at the end of the treatment | up to 24 weeks

OTHER OUTCOMES:
MR Imaging changes of orbital contents compared with the baseline after 4 times and at the end of the treatment | up to 24 weeks
  Including: exophthalmos, the volume of the lacrimal gland/optic nerve/extraocular muscle/retroorbital adipose tissue/lacrimal gland, edema, inflammation, blood perfusion, fibrosis, and fatty changes
Percentage of participants who underwent surgery throughout the study period | throughout the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided